CLINICAL TRIAL: NCT06147830
Title: A Multinational Observational Longitudinal Study to Describe the Patient Characteristics, Health Care Interventions, and Health Outcomes of Patients With Major Bleedings in the Presence of Factor Xa Inhibitor Treatment
Brief Title: A Study to Describe the Characteristics, Health Care Interventions and Outcomes of Patients With Major Bleedings in the Presence of Factor Xa Inhibitor Treatment
Acronym: REVERXaL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D9603R00003
Record Dates: First submitted 2023-10-23; First posted 2023-11-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Major Bleeding
Keywords: real-world evidence; Factor Xa inhibitor treatment; reversal/replacement therapy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A - Historical Cohort: Cohort A will comprise of approximately 2000 patients admitted for major bleedings in the presence of Factor Xa inhibitor treatment during a defined period (up to 2 years prior to commencing enrolment of patients in Cohort B). Patients who developed major bleeding in the presence of Factor Xa inhibitor treatment while already admitted in hospitals will also be included. Patients may or may not have received a reversal/replacement therapy. Patients are followed in medical charts from admission to discharge.
  Interventions: Other: None (Observational study)
- Cohort B - Prospective Cohort: Cohort B will enrol approximately 2000 patients who were administered any reversal or replacement agent during the acute care phase for a major bleeding in the presence of Factor Xa inhibitor treatment at the participating sites. Patients will be followed up to three months after administration of reversal or replacement therapy.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — Not Applicable since Observational Study
  Other Names: Observational Study

SUMMARY:
REVERXaL study aims to increase the understanding of the patient characteristics, bleeding presentation, health care interventions provided, and the clinical as well as self-reported health outcomes of patients with major bleeding in the presence of Factor Xa inhibitor treatment. The generation of insight on treatment approaches and associated outcomes in hospitalized patients with Factor Xa inhibitor-related major bleeds may inform clinical guidelines, health system decision making and streamline treatment pathways in this population.

DETAILED DESCRIPTION:
REVERXaL is a multinational observational study incorporating 2 patient cohorts (historical and prospective) with major bleeds during Factor Xa inhibitor use. This study will be mainly descriptive in nature without any pre-specified statistical hypotheses. Variables will be collected according to routine medical practice either through primary data collection directly from patients, or from secondary data collection via data extraction from electronic or paper medical records into electronic case report forms (eCRFs). Patients will undergo clinical assessments and receive standard medical care as determined by their treating physicians. Patients will not receive any experimental disease management intervention or experimental treatment because of their participation in the study. As part of routine care, study investigators will evaluate patients about their medical history, medication history, bleeding presentation, and any adverse event (AE) or severe adverse event (SAE) experiences since the previous clinical visit and the related information. No additional or pre-defined site visits will be scheduled outside of the patient's routine clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years on the index date
* Admitted to the hospital with an acute major bleeding or developed an acute bleeding while already in hospital
* Ongoing treatment with a Factor Xa inhibitor before the index date
* Provided signed and dated informed consent or able to obtain a waiver

In addition, for cohort B:

- Administered reversal or replacement therapy

Exclusion Criteria:

* Pregnant women
* Patients enrolled in any interventional trial that includes reversal/replacement agents

In addition, for cohort B:

* Use of vitamin K antagonists, dabigatran, prothrombin complex concentrates or recombinant factor VII, or transfusion of whole blood or plasma within the preceding 7 days of the index event
* As judged by the investigator, if it is deemed undesirable for the patient to participate in the study or participant is unlikely to comply with study procedures, and requirements
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥18 years admitted to hospital with an acute major bleeding or developed an acute bleeding while already in hospital and received ongoing treatment with a Factor Xa inhibitor before the index date.
Sampling Method: Non-Probability Sample
Enrollment: 2202 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Demographics (age in years) | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  Summary statistics will be used to describe demographics.
Demographics (sex) | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  Summary statistics will be used to describe demographics.
Demographics (ethnicity) | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  Summary statistics will be used to describe demographics.
Demographics (race) | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  Summary statistics will be used to describe demographics.
Demographics (payer type) | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  Summary statistics will be used to describe demographics.
Clinical presentation | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  Summary statistics will be used to describe clinical presentation of patients.
Healthcare interventions provided during acute care phase | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  To describe the health care interventions provided during acute care phase in patients with major bleedings in the context of Factor Xa inhibitor treatment.
In-hospital outcomes | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  To describe the in-hospital outcomes in patients with major bleedings in the context of Factor Xa inhibitor treatment.
Timing of administration of reversal/replacement agents since admission/bleed onset | Cohort A: from admission for the bleeding (index date) until hospital discharge. Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  To describe the timing of administration of reversal/replacement agents from admission/bleed onset.
Short Form Health Survey (SF-36) - Cohort B | Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  The 36-Item Short Form Health Survey Version 2 (SF-36 v2) is a standardized, patient-administered instrument across eight domains (including physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health). Each subscale is scored separately, and the scores range from 0 to 100. Higher scores indicate better health-related quality of life.
5-Dimension Health Questionnaire 5 Level (EQ-5D-5L) - Cohort B | Cohort B: from index date (time of administration of reversal/replacement agent) to hospital discharge (up to 90 days)
  The EuroQoL EQ-5D-5L questionnaire measures generic Health-Related Quality of Life (HRQoL) and contains questions on five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety/depression. Each subscale is scored based on 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). It can be converted into a single numeric score and has been translated and validated in numerous countries. The EQ-5D-5L scoring system assigns a utility value to each health state based on population preferences. The utility values range from -0.594 (representing the worst health state possible) to 1.000 (representing perfect health).

SECONDARY OUTCOMES:
Clinical outcomes - Cohort B | At 30 days post index (date of administration of reversal/replacement agents)
  To describe the clinical outcomes in patients who experienced major bleedings in the context of Factor Xa inhibitor treatment and administered reversal/replacement therapy.
Timing of administration of reversal/replacement therapy since admission/bleed onset - Cohort B | At 30 days post index (date of administration of reversal/replacement agents)
  To describe the timing of administration of reversal replacement therapy since admission/bleed onset.
Short Form Health Survey (SF-36) - Cohort B | 30 days post index (date of administration of reversal/replacement agents)
  The 36-Item Short Form Health Survey Version 2 (SF-36 v2) is a standardized, patient-administered instrument across eight domains (including physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Each subscale is scored separately, and the scores range from 0 to 100. Higher scores indicate better health-related quality of life.
5-Dimension Health Questionnaire 5 Level (EQ-5D-5L) - Cohort B | 30 days post index (date of administration of reversal/replacement agents)
  The EuroQoL EQ-5D-5L questionnaire measures generic HRQoL and contains questions on five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety/depression. Each subscale is scored based on 5 levels of severity (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). It can be converted into a single numeric score and has been translated and validated in numerous countries. The EQ-5D-5L scoring system assigns a utility value to each health state based on population preferences. The utility values range from -0.594 (representing the worst health state possible) to 1.000 (representing perfect health).

CONTACTS AND LOCATIONS:
Locations (75):
- United States (25):
  - Research Site, Chandler, Arizona
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, Torrance, California
  - Research Site, Lakewood, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Glenview, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Royal Oak, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Albany, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Staten Island, New York
  - Research Site, Stony Brook, New York
  - Research Site, Valhalla, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Research Site, Milwaukee, Wisconsin
- Germany (22):
  - Research Site, Aachen
  - Research Site, Altenburg
  - Research Site, Bad Neustadt/Saale
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, G Ppingen
  - Research Site, Jena
  - Research Site, Koblenz
  - Research Site, L Beck
  - Research Site, L Neburg
  - Research Site, Leipzig
  - Research Site, Ludwigshafen am Rhein
  - Research Site, Osnabr Ck
  - Research Site, Potsdam
  - Research Site, Trier
  - Research Site, Tübingen
  - Research Site, Würzburg
- Japan (16):
  - Research Site, Asahikawa
  - Research Site, Fukuoka
  - Research Site, Hitachi
  - Research Site, Izumo
  - Research Site, Kagoshima
  - Research Site, Kamakura
  - Research Site, Kitakyushu
  - Research Site, Kyoto
  - Research Site, Mitaka
  - Research Site, Nagakute
  - Research Site, Okayama
  - Research Site, Saga
  - Research Site, Shimotsuke
  - Research Site, Suita
  - Research Site, Tachikawa
  - Research Site, Tokyo
- United Kingdom (12):
  - Research Site, Aberdeen
  - Research Site, Bournemouth
  - Research Site, Canterbury
  - Research Site, Cardiff
  - Research Site, Edgbaston
  - Research Site, Harrow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Preston
  - Research Site, Sheffield
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Alikhan R, Nour M, Yasaka M, Ofori-Asenso R, Axelsson-Cheramy S, Chen H, Seghal V, Yokobori S, Koch B, Tiede A, Cash BD, Maegele M, Singer AJ. Design and rationale for REVERXaL: A real-world study of patients with factor Xa inhibitor-associated major bleeds. Thromb Res. 2024 Aug;240:109046. doi: 10.1016/j.thromres.2024.109046. Epub 2024 Jun 5. PMID 38905928
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9603R00003&attachmentIdentifier=aaf79989-4c6c-4fed-bf4f-1394c039598c&fileName=d9603r00003_Redacted_CSR_synopsis.pdf&versionIdentifier=